CLINICAL TRIAL: NCT06573645
Title: A Phase III Randomized Controlled Study Comparing High-dose Rituximab (500 mg/m²) Combined With CHOP Regimen Versus Standard-dose Rituximab (375 mg/m²) Combined With CHOP Regimen in Male Patients With Newly Diagnosed Advanced Diffuse Large B-cell Lymphoma
Brief Title: A Phase III Clinical Trial of High-dose Rituximab (500mg/m²) Combined With CHOP Regimen in the Treatment of Male Patient With Newly Diagnosed Advanced DLBCL
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xia Yi (Other)
Responsible Party: Sponsor-Investigator, Xia Yi, Director, Sun Yet-Sen University Cancer Center
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-380
Record Dates: First submitted 2024-08-02; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: lymphoma; Diffuse large B cell lymphoma; High doses rituximab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: A non-repetitive stratified block randomization method is used, with the treatment assignment codes for participants (randomization table) being generated by a blinded statistician in a 1:1 ratio. The randomization table is then uploaded to the central randomization system for configuration. Once a participant's eligibility is confirmed, the researcher logs into the central randomization system, enters the participant's information, and obtains the participant's random number and drug code. The researcher administers the corresponding study treatment based on the drug code. Participants are randomized in a 1:1 ratio to either the experimental group (rituximab 500 mg/m²) or the control group (rituximab 375 mg/m²).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose Rituximab Group (Experimental): Patients will be assigned to the trial group (rituximab 500 mg/m2) and will receive six cycles of R-CHOP (21 days per cycle), followed by two maintenance cycles of rituximab (21 days per cycle).
  Interventions: Drug: Rituximab
- Standard-dose Rituximab Group (Active Comparator): Patients will be assigned to the control group (rituxan 375 mg/m2), the participants will receive 6 cycles R - CHOP treatment (21 d for a cycle), and the subsequent 2 cycle rituxan maintenance therapy (21 d for a cycle)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Patients will be randomized to receive either rituximab 500 mg/m2 or rituximab 375 mg/m2 for six cycles of R-CHOP (21 days per cycle), followed by two maintenance cycles of rituximab (21 days per cycle).

SUMMARY:
Comparison of MODIFIED progression-free survival (Modified-PFS) in high-dose rituximab (500mg/m²) plus CHOP versus standard-dose rituximab plus CHOP in previously untreated (TN) stage III-IV male DLBCL patients

DETAILED DESCRIPTION:
This study is a multicenter, randomized, controlled Phase III clinical trial that primarily evaluates the modified progression-free survival (MODIFIED-PFS) in previously untreated male DLBCL patients treated with high-dose rituximab (500mg/m²) combined with the CHOP regimen compared to standard-dose rituximab combined with the CHOP regimen. After signing the informed consent and before randomization, all participants must provide sufficient tumor tissue biopsy samples for confirmation of DLBCL via central laboratory tests such as HE staining and IHC. Eligible participants are randomized in a 1:1 ratio to either the experimental group (rituximab 500 mg/m2) or the control group (rituximab 375 mg/m2) and will receive 6 cycles of R-CHOP treatment (21 days per cycle), followed by 2 additional cycles of maintenance therapy with rituximab (21 days per cycle).

ELIGIBILITY:
Key Inclusion Criteria:

1. age <75y, male patients
2. According to the 2017 Revised WHO Classification criteria for lymphoma, the subject was diagnosed with DLBCL
3. According to Ann Arbor staging, patients were classified as stage III-IV patients
4. No previous anti-tumor systemic therapy or local radiation therapy for DLBCL
5. Expected survival ≥6 months
6. Have sufficient coagulation function and liver and kidney function
7. Haver sufficient bone marrow function
8. All patients should take medically approved contraceptive measures within 12 months after rituximab administration (specific circumstances should follow the listed drug label)
9. Subjects were enrolled voluntarily, signed informed consent, and followed the experimental treatment protocol and visit plan

Key Exclusion Criteria:

1. Subjects assessed by the investigator to be intolerant to the R-CHOP regimen and/or any drug therapy;
2. Any previous anti-lymphoma systemic therapy or local radiation therapy
3. Consider patients with lymphoma involving the central nervous system (CNS) or diagnosed with primary CNS lymphoma (PCNSL); The diagnosis was primary mediastinal large B-cell lymphoma (PMBL)
4. Previously received organ transplantation or hematopoietic stem cell transplantation
5. Had received major surgery or major trauma within 4 weeks before the first medication (or before randomization), and had participated in clinical trials of non-anti-tumor drugs or medical devices within 4 weeks
6. Have had malignant tumors other than the indications targeted in this study in the past three years
7. Participants with any serious and/or uncontrolled systemic disease who are determined by the investigator to be unsuitable for participation in the study
8. Major cardiovascular disease occurred within 6 months before the first medication (or before randomization)
9. Any conditions that affect the patient's ingestion of the drug, as well as conditions that seriously affect the absorption or pharmacokinetic parameters of the drug in the trial, including difficult to control nausea and vomiting, short bowel syndrome, etc.
10. Subjects who received live or attenuated vaccine within 4 weeks prior to initial administration (or prior to randomization) or planned to receive live vaccine during the study period or 4 weeks after the end of study treatment
11. A hemorrhagic disease (such as von Willebrand disease or hemophilia A, hemophilia B, etc.) or according to the judgment of the investigator has a clear bleeding tendency
12. have a serious peripheral nervous system or central nervous system disease.
13. Warfarin or other vitamin K antagonists are required during the study
14. There is an autoimmune disease that cannot be controlled or requires treatment within 4 weeks prior to the first dose (or prior to randomization)
15. Doxorubicin has been used in the past ≥150 mg/m2
16. The investigator believes that the subjects have other conditions that are not suitable for participation in this experiment.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 428 (Estimated)
Dates: Start 2024-08-23 (Estimated); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-07-12 (Estimated)

PRIMARY OUTCOMES:
MODIFIED-PFS | From the date of enrollment until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  To investigate the preliminary anti-tumor efficacy

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of enrollment until the date of death from ant cause, assessed up to 48 months
  To investigate the preliminary anti-tumor efficacy
Complete response rate (CRR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy
Objective response rate (ORR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-07-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT06573645/Prot_000.pdf
  • Informed Consent Form (2024-07-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT06573645/ICF_001.pdf